CLINICAL TRIAL: NCT00065390
Title: Pilot (Phase I-II) Study of Pyrimethamine (Daraprim) for the Treatment of the Autoimmune Lymphoproliferative Syndrome (ALPS)
Brief Title: Pyrimethamine to Treat Autoimmune Lymphoproliferative Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030248; 03-I-0248
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-06

CONDITIONS: Autoimmune Disease; Lymphatic Disease; Lymphoproliferative Disorder
Keywords: ALPS; Pyrimethamine; Folinic Acid; Lymphadenopathy; Splenomegaly; Autoimmune Lymphoproliferative Syndrome
MeSH Terms: conditions — Autoimmune Diseases; Lymphatic Diseases; Lymphoproliferative Disorders; Lymphadenopathy; Splenomegaly; Autoimmune Lymphoproliferative Syndrome | interventions — Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine

SUMMARY:
This study will examine whether the drug pyrimethamine can shrink lymph nodes and spleen in patients with autoimmune lymphoproliferative syndrome (ALPS). In this disease, lymphocytes (white blood cells) do not die as they normally would. As a result, patients have enlarged lymph glands, spleen, or liver, and other problems that may involve blood cell counts and autoimmune disease (overactivity of the immune system). Pyrimethamine is an orally administered antibiotic that has been used to treat or prevent malaria and toxoplasma, and may be effective in shrinking lymph nodes and spleen.

Patients with ALPS who are between 2 and 70 years of age and have had lymph gland enlargement for at least 1 year may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, and possibly a bone marrow test. Females of reproductive age will be screened with a urine pregnancy test. Women who are capable of becoming pregnant must use an effective method of birth control during the entire study period, because, taken during early months of pregnancy, pyrimethamine can cause birth defects in the fetus. Women who are pregnant or nursing are excluded from the study.

Participants will undergo the following tests and procedures:

* CT scan: For this test, the patient lies still in the CT scanner while images are taken of the neck, chest, and stomach area. A contrast dye is injected into a vein to brighten the CT images. Very young children will be evaluated on a case by case basis to determine whether a CT scan will be performed.
* Bone marrow biopsy: Participants undergo this test to rule out underlying bone marrow disease if they have not had a bone marrow test done in the last six months prior to enrolling in pyrimethamine study, as pyrimethamine can affect bone marrow function. Under local anesthesia, a needle is inserted into the back part of the hipbone and a small amount of marrow is removed. (Children are sedated for this test.)
* Leukapheresis: This is a procedure for collecting a small proportion of circulating white blood cells while conserving the majority of blood cells. Specifically, blood is drawn from a needle placed in an arm vein and is directed into a cell separator machine, which separates the blood cells by spinning. A small proportion of circulating white cells are removed, and the red cells, platelets, plasma and majority of white cells are returned to the patient's blood circulation. Only patients who are 7 years of age or older and weigh at least 55 pounds undergo this procedure. Other participants who choose not to have apheresis will have about 3 tablespoons of blood drawn instead.
* Pyrimethamine administration: When the above tests are completed, participants begin taking pyrimethamine. The dose is determined according to the individual's weight and is gradually increased during the study period. Patients take the drug twice a week for a total of 12 weeks.
* Blood tests: Blood samples are collected during weeks 2, 4, 6, 8, and 10 after beginning treatment, and 2 weeks after the last dose of pyrimethamine. The purpose of these blood tests is to check for possible drug-related side effects. Patients who develop a skin rash, mouth sores or other side effects may have one or more doses of the treatment drug withheld. When indicated, the patient will be directed to stop taking the study drug. If needed, drug side effects will be treated with a vitamin supplement, folinic acid, taken by mouth, 3 times weekly.
* Evaluations at the NIH Clinical Center will comprise of a pretreatment visit, one end of treatment visit at the end of 12 weeks and an optional post-treatment visit 3months after stopping pyrimethamine therapy.

Patients who respond well to treatment may be asked to return to NIH for additional visits at 3, 6, and 12 months after the treatment has ended for repeat evaluations. If their lymph glands or spleen become much larger after stopping pyrimethamine, they will be offered treatment for another 12 weeks. If they respond to the second course of treatment, they will return to NIH again after 3, 6, and 12 months. If the symptoms return again, patients will be asked to resume treatment for an additional 6 months or more. They will have blood drawn periodically by their private physician and will return to NIH for evaluation every 12 weeks.

DETAILED DESCRIPTION:
The Autoimmune Lymphoproliferative Syndrome (ALPS) is an inherited disease associated with a defect of lymphocyte apoptosis that leads to lymphoproliferation and autoimmunity. Although, there are treatments for many of its complications, there currently is no safe and effective therapy for this syndrome itself. Recently investigators in Europe serendipitously observed that some children with ALPS showed reductions in spleen and lymph node size while in pyrimethamine/sulfadoxine (Fansidar) for Pneumocystis carinii prophylaxis. Our own subsequent pilot clinical trial of Fansidar (Protocol #01-I-0132) was terminated after failure to recruit well-defined ALPS patients who lacked histories suspicious for allergies to sulfa drugs. Our own in vitro studies, however revealed that pyrimethamine and not sulfadoxine induces lymphocyte apoptosis and this observation has suggested to us that pyrimethamine may be beneficial alone, thus avoiding the added risks of allergy and hypersensitivity associated with the sulfa drugs. However, potential bone marrow toxicity that may result from an escalating dose schedule of pyrimethamine should respond to the addition of folinic acid (Leucovorin) to the regimen.

We propose to conduct a pilot study on the safety and efficacy of the drug, pyrimethamine for the treatment of ALPS. Six to 8 individuals, with ALPS will be treated for up to 3 months, initially, with twice-weekly pyrimethamine (Daraprim) at escalating doses adjusted by weight, with the addition of folinic acid when needed to aid management of marrow toxicity. The effects of pyrimethamine treatment on lymph node and/or spleen size will be assessed by CT scan. The effect of treatment on other laboratory features of ALPS will also be assessed. Evaluating the effects of pyrimethamine on these clinical and laboratory parameters will allow us to determine if this drug demonstrates sufficient activity to warrant study in a larger randomized controlled trial.

ELIGIBILITY:
INCLUSION CRITERIA:

All subjects must fulfill the published criteria for the diagnosis of ALPS (documented nonmalignant lymphadenopathy and/or splenomegaly of at least 1 year duration; greater than or equal to 1% TCR alpha/beta(+) CD4(-)CD8(-) T cells in the peripheral blood and defective apoptosis by in vitro assay). This must include clinically documented lymphadenopathy involving more than two nodes in more than one regional group of nodes measuring greater than 1 cm in size and/or a palpable spleen.

Age greater than 2 years and less than 70 years.

Must have a personal primary care physician.

Women of reproductive age and potential must have a negative pregnancy test at study entry and commit to using an acceptable method of barrier or hormonal contraception (e.g. condoms, diaphragms, oral contraceptives and long acting progestin agents) if sexually active during the study and for 3 months after the last dose of pyrimethamine.

Must be willing to sign a consent form.

EXCLUSION CRITERIA:

Patient will be excluded if any of the following is present:

Weight of less than 10 kilograms (22 lbs).

Patients receiving and requiring anti-folate drugs such as sulfonamides, trimethoprim, pyrimethamine and methotrexate for any other purpose. They should be off these medications, including Bactrim, for at least 7 days prior to enrolling in this protocol.

Megaloblastic anemia, folate deficiency or a mean corpuscular volume greater than 125 in last three months with evidence of megaloblastic changes in the bone marrow.

A hemoglobin concentration of less than 8 gm/dl, a platelet count of less than 50 K/mm(3), or an absolute neutrophil count of less than 500/mm(3), at study entry or during the study period.

Liver disease determined by an ALT, AST or bilirubin 3 times above the upper limit of normal.

Renal dysfunction determined by a calculated urine creatinine clearance of less than or equal to 70 ml/min/1.73 m(2) in children and less than or equal to 60 ml/min in adults or using the Schwartz formula or Levy formula based on serum creatinine.

Patients on immunosuppression (eg: corticosteroid, azathioprine, cyclosphosphamide, etc) are eligible if the dose of the immunosuppressive drug has been stable for at least 3 months prior to enrollment and their hematologic parameters meet the criteria outlined in item 4 (above).

Pregnancy. Women of reproductive age and potential must have a negative pregnancy test at study entry and commit to using an acceptable method of barrier or hormonal contraception (e.g. condoms, diaphragms, oral contraceptives and long acting progestin agents) if sexually active during the study and for 3 months after the last dose of pyrimethamine.

Lactating mothers who are breast feeding their babies will not be eligible.

ALPS patients who have been treated with bone marrow toxic chemotherapy regimens for Hodgkins and Non-Hodgkins lymphoma or other malignancies are not eligible for this pilot study.

Unwilling or unable to comply with the need to have periodic blood tests to monitor possible side effects of treatment, or other major requirements of this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 2003-07; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sneller MC, Wang J, Dale JK, Strober W, Middelton LA, Choi Y, Fleisher TA, Lim MS, Jaffe ES, Puck JM, Lenardo MJ, Straus SE. Clincal, immunologic, and genetic features of an autoimmune lymphoproliferative syndrome associated with abnormal lymphocyte apoptosis. Blood. 1997 Feb 15;89(4):1341-8. PMID 9028957
- [Background] Straus SE, Sneller M, Lenardo MJ, Puck JM, Strober W. An inherited disorder of lymphocyte apoptosis: the autoimmune lymphoproliferative syndrome. Ann Intern Med. 1999 Apr 6;130(7):591-601. doi: 10.7326/0003-4819-130-7-199904060-00020. PMID 10189330
- [Background] Avila NA, Dwyer AJ, Dale JK, Lopatin UA, Sneller MC, Jaffe ES, Puck JM, Straus SE. Autoimmune lymphoproliferative syndrome: a syndrome associated with inherited genetic defects that impair lymphocytic apoptosis--CT and US features. Radiology. 1999 Jul;212(1):257-63. doi: 10.1148/radiology.212.1.r99jl40257. PMID 10405750